CLINICAL TRIAL: NCT01371630
Title: Phase I/II Study of the Combination of Inotuzumab Ozogamycin (CMC-544) With Low-Intensity Chemotherapy in Patients With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Inotuzumab Ozogamicin and Combination Chemotherapy in Treating Patients With Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0991; NCI-2011-01123 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0991 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative; Burkitt-Like Lymphoma With 11q Aberration; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; Recurrent B Acute Lymphoblastic Leukemia; Recurrent Burkitt Lymphoma; Refractory B Acute Lymphoblastic Leukemia; Refractory Burkitt Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab; Cyclophosphamide; Cytarabine; Dexamethasone; Inotuzumab Ozogamicin; Mercaptopurine; Methotrexate; Prednisone; Rituximab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (inotuzumab ozogamicin, combination chemotherapy) (Experimental): See Detailed Description Arm I
  Interventions: Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Biological: Inotuzumab Ozogamicin; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine
- Arm II (inotuzumab ozogamicin, combination chemotherapy) (Experimental): See Detailed Description Arm II
  Interventions: Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Biological: Inotuzumab Ozogamicin; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine
- Arm III (inotuzumab ozogamicin, combination chemotherapy) (Experimental): See Detailed Description Arm III
  Interventions: Biological: Blinatumomab; Drug: Cytarabine; Drug: Dexamethasone; Biological: Inotuzumab Ozogamicin; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Biological: Rituximab; Drug: Vincristine

INTERVENTIONS:
Biological: Blinatumomab — Given CIVI
Drug: Cyclophosphamide — Given IV
  Arms: Arm I (inotuzumab ozogamicin, combination chemotherapy); Arm II (inotuzumab ozogamicin, combination chemotherapy)
Drug: Cytarabine — Given IT and IV
Drug: Dexamethasone — Given IV or PO
Biological: Inotuzumab Ozogamicin — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mercaptopurine — Given PO
  Arms: Arm I (inotuzumab ozogamicin, combination chemotherapy); Arm II (inotuzumab ozogamicin, combination chemotherapy)
Drug: Methotrexate — Given IT, IV, and PO
Drug: Prednisone — Given PO
  Arms: Arm I (inotuzumab ozogamicin, combination chemotherapy); Arm II (inotuzumab ozogamicin, combination chemotherapy)
Biological: Rituximab — Given IV
Drug: Vincristine — Given IV

SUMMARY:
This phase I/II trial studies the side effects and best dose of inotuzumab ozogamicin and to see how well it works when given together with combination chemotherapy in treating patients with acute lymphoblastic leukemia. Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a toxic agent called N-acetyl-gamma-calicheamicin dimethyl hydrazide (CalichDMH). Inotuzumab attaches to CD22 positive cancer cells in a targeted way and delivers CalichDMH to kill them. Immunotherapy with monoclonal antibodies, such as blinatumomab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving inotuzumab ozogamicin together with combination chemotherapy may be a better treatment for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of inotuzumab ozogamicin (inotuzumab ozogamycin) in combination with low-intensity chemotherapy in elderly patients (age 60 or older) with acute lymphoblastic leukemia (ALL). (Phase I)

II. Evaluate the efficacy of inotuzumab ozogamycin in combination with low-intensity chemotherapy in elderly and unfit to receive intensive therapy patients with ALL. (Phase II)

III. To evaluate the side effects of the treatment. (Phase II)

IV. Evaluate the regimen efficacy in refractory-relapsed ALL. (Phase II)

EXPLORATORY OBJECTIVES:

I. To identify genomic alterations in adult ALL predictive for response and long-term outcomes with the combination of hyper-CVD (cyclophosphamide, dexamethasone, methotrexate, and cytarabine) + inotuzumab + blinatumomab.

II. To evaluate the impact of next generation sequencing (NGS)-based minimal residual disease (MRD) assay on outcomes and to compare with standard flow cytometry MRD assays.

OUTLINE: This is a phase I, dose-escalation study of inotuzumab ozogamicin followed by a phase II study. Patients are assigned to 1 of 3 arms.

ARM I (UNTREATED):

CYCLES 1, 3, 7, AND 9: Patients receive cyclophosphamide intravenously (IV) over approximately 3 hours twice daily (BID) on days 1-3; vincristine IV over 30 minutes on days 1 and 8; dexamethasone IV or orally (PO) on days 1-4 and 11-14; inotuzumab ozogamicin IV over approximately 1 hour on day 3 of cycle 1 and day 2 or 3 of cycle 3; methotrexate intrathecally (IT) on day 2 of cycles 1 and 3; and cytarabine IT on day 8 of cycles 1 and 3. Patients may also receive rituximab IV on days 1 and 8 of cycles 1 and 3. Cycles alternate every 3-4 weeks in the absence of disease progression or unacceptable toxicity.

CYCLES 2, 4, 8, AND 10: Patients receive methotrexate IV over approximately 2 hours and then continuously over approximately 22 hours on day 1; cytarabine IV over approximately 3 hours BID on days 2-3; inotuzumab ozogamicin IV over approximately 1 hour on day 2 or 3 of cycles 2 and 4; cytarabine IT on day 5 of cycles 2 and 4; and methotrexate IT on day 8 of cycles 2 and 4. Patients may also receive rituximab IV on days 1 and 8 of cycles 2 and 4. Cycles alternate every 3-4 weeks in the absence of disease progression or unacceptable toxicity.

CYCLES 5-8: Patients receive blinatumomab as a continuous intravenous infusion (CIVI) on days 1-29. Patients also receive dexamethasone IV over 15-30 minutes on day 1 and 3 of cycle 5 and then day 1 of cycles 6-8. Treatment repeats every 42 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive mercaptopurine PO BID and methotrexate PO once weekly for 3 years. Patients also receive vincristine IV over 30 minutes once monthly and prednisone PO daily five times a month for 1 year. Patients receive blinatumomab CIVI on days 1-28 of cycles 4, 8, 12, and 16. Cycles repeat every 42 days for 3 years in the absence of disease progression or unacceptable toxicity.

ARM II (RELAPSED/REFRACTORY):

CYCLES 1, 3, AND 5: Patients receive cyclophosphamide IV over approximately 3 hours BID on days 1-3; vincristine IV over 30 minutes on day 1; rituximab IV over 2-6 hours on days 1 and 8 of cycles 1 and 3; dexamethasone IV or PO on days 1-4; inotuzumab ozogamicin IV over 1 hour on days 2 and 8; methotrexate IT on day 2 of cycles 1 and 3; cytarabine IT on day 8 of cycles 1 and 3; and blinatumomab CIVI on days 4-21. Cycles alternate every 4 weeks in the absence of disease progression or unacceptable toxicity.

CYCLES 2, 4, AND 6: Patients receive methotrexate IV over 24 hours on day 1; cytarabine IV over approximately 3 hours BID on days 2-3; rituximab IV over 2-6 hours on days 1 and 8 of cycles 2 and 4; inotuzumab ozogamicin IV over 1 hour on days 2 and 8 of cycles 2 and 4; cytarabine IT on day 2 of cycles 2 and 4, methotrexate IT on day 8 of cycles 2 and 4; and blinatumomab CIVI on days 4-21. Cycles alternate every 4 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive mercaptopurine PO BID and methotrexate PO once weekly for 3 years. Patients also receive vincristine IV over 30 minutes once monthly and prednisone PO daily five times a month for 1 year. Patients receive blinatumomab CIVI on days 1-28 of cycles 4, 8, 12, and 16. Cycles repeat every 42 days for 3 years in the absence of disease progression or unacceptable toxicity.

ARM III (70 YEARS AND OLDER):

INDUCTION CYCLE (CYCLE 1): Patients receive dexamethasone IV or PO on days 1-4; vincristine IV over 30 minutes on day 1; inotuzumab ozogamicin IV over 1 hour on days 1 and 8 of cycle 1; blinatumomab CIVI on days 15-28. Patients may also receive rituximab IV on days 2 and 9.

INTRATHECAL PROPHYLAXIS: Patients receive methotrexate IT alternating with cytarabine IT on days 2 and 8 of cycles 1 and 3, and cytarabine IT alternating with methotrexate IT on days 2 and 8 of cycles 2 and 4. Treatment repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION (CYCLES 2-5): Patients receive blinatumomab CIVI on days 1-28; inotuzumab ozogamicin IV over 1 hour on days 1 and 8 of cycles 2-4. Patients may also receive rituximab IV on days 2 and 9 of cycles 2-4. Treatment repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 60 years or older with previously untreated ALL pre-B, Philadelphia chromosome (Ph-) negative or (Ph+) positive ALL Minimal prior therapy (less than 1 week of steroids, vincristine, and/or 1 dose of anthracycline or alkylating agents) are allowed.
2. Patients unfit ≥ 18 - < 60 years of age with previously untreated ALL pre- B, Philadelphia chromosome (Ph-) negative or (Ph+) positive ALL (includes patients initiated on first cycle of hyper-CVAD before cytogenetics known. These patients could have received one or two cycles of chemotherapy with or without other TKIs and still eligible.

   These patients are defined as having at least one of the below comorbidities:
   1. ECOG performance status ≥ 2
   2. Severe cardiac disorder (e.g., congestive heart failure requiring treatment, ejection fraction ≤ 50%, or chronic stable angina)
   3. Severe pulmonary disorder (e.g., DLCO ≤ 65% or FEV1 ≤ 65%)
   4. Creatinine clearance < 45 mL/min, and
   5. Hepatic disorder with total bilirubin > 1.5 x upper limit of normal

   <!-- -->

   1. If they achieved CR, they are assessable only for event-free and overall survival, or
   2. If they failed to achieve CR, they are assessable for CR, event-free, and overall survival
3. Patients age 60 years and older unfit for intensive chemotherapy with one or more comorbidities (e.g., renal insufficiency, heart disease, cardio-vascular disease, uncontrolled hypertension, diabetes, respiratory problems, among others) and a PS of ≥ 1. All ages of Jehovah's witness are eligible.
4. Zubrod performance status 0-3.
5. Adequate liver function (bilirubin < 1.95 mg/dL and SGPT or SGOT < 3 x upper limit of normal [ULN], unless considered due to tumor), and renal function (estimated creatinine clearance ≥50 mL/min/1.73 m2). Even if organ function abnormalities are considered due to tumor, the upper limit for bilirubin is < 2.6 mg/dL and creatinine < 3 mg/dL.
6. Provision of written informed consent.
7. Patients in first remission are eligible.
8. Patients with refractory-relapsed ALL, Burkitt lymphoma, Burkitt-like lymphoma with 11q aberration, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, and high-grade B-cell lymphoma not otherwise specified with marrow involvementBof any age are eligible.

Exclusion Criteria:

1. Newly diagnosed Burkitt's Leukemia or Lymphoma, T-cell ALL or lymphoblastic lymphoma.
2. Patient with active heart disease (NYHA class > 3 as assessed by history and physical examination).
3. Patients with a cardiac ejection fraction (as measured by either MUGA or echocardiogram) < 40% are excluded.
4. Patients with active hepatitis are excluded.
5. Pregnant or breast-feeding women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2011-08-26 (Actual); Primary Completion 2027-12-25 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of inotuzumab ozogamicin based on incidence of dose limiting toxicities (Phase I) | 28 days
  Defined as non-hematologic grade 3 or 4 toxicities during the first course. Toxicities will be monitored using the method of Thall, Simon, and Estey. Adverse events will be summarized and toxicity rate will be estimated with a 90% credible interval.
Progression free survival (PFS) in frontline elderly acute lymphoblastic leukemia (ALL) (Phase II) | 2 years
  Bayesian time-to-event model will be used. Kaplan and Meier product limit method will be used to estimate the PFS along with the 95% confidence intervals for the median PFS. Univariate and multivariate Cox proportional hazards regression models will be used to identify prognostic factors.
Response rate in refractory-relapsed acute lymphoblastic leukemia (ALL) (Phase II) | Up to 5 years
  The precise complete remission (CR) and marrow CR rate will be defined.
Survival in refractory-relapsed acute lymphoblastic leukemia (ALL) (Phase II) | Up to 1 year
  The median and 1-year survival rate will be defined. Kaplan and Meier product limit method will be used to estimate the overall survival (OS) along with the 95% confidence intervals for the median OS. Univariate and multivariate Cox proportional hazards regression models will be used to identify prognostic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Zhao Y, Short NJ, Kantarjian HM, Chang TC, Ghate PS, Qu C, Macaron W, Jain N, Thakral B, Phillips AH, Khoury J, Garcia-Manero G, Zhang W, Fan Y, Yang H, Garris RS, Nasr LF, Kriwacki RW, Roberts KG, Konopleva M, Jabbour EJ, Mullighan CG. Genomic determinants of response and resistance to inotuzumab ozogamicin in B-cell ALL. Blood. 2024 Jul 4;144(1):61-73. doi: 10.1182/blood.2024023930. PMID 38551807
- [Derived] Jabbour E, Short NJ, Senapati J, Jain N, Huang X, Daver N, DiNardo CD, Pemmaraju N, Wierda W, Garcia-Manero G, Montalban Bravo G, Sasaki K, Kadia TM, Khoury J, Wang SA, Haddad FG, Jacob J, Garris R, Ravandi F, Kantarjian HM. Mini-hyper-CVD plus inotuzumab ozogamicin, with or without blinatumomab, in the subgroup of older patients with newly diagnosed Philadelphia chromosome-negative B-cell acute lymphocytic leukaemia: long-term results of an open-label phase 2 trial. Lancet Haematol. 2023 Jun;10(6):e433-e444. doi: 10.1016/S2352-3026(23)00073-X. Epub 2023 May 12. PMID 37187201
- [Derived] Kantarjian H, Haddad FG, Jain N, Sasaki K, Short NJ, Loghavi S, Kanagal-Shamanna R, Jorgensen J, Khouri I, Kebriaei P, Alvarado Y, Kadia T, Paul S, Garcia-Manero G, Dabaja B, Yilmaz M, Jacob J, Garris R, O'Brien S, Ravandi F, Jabbour E. Results of salvage therapy with mini-hyper-CVD and inotuzumab ozogamicin with or without blinatumomab in pre-B acute lymphoblastic leukemia. J Hematol Oncol. 2023 May 2;16(1):44. doi: 10.1186/s13045-023-01444-2. PMID 37131217
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] Kantarjian H, Ravandi F, Short NJ, Huang X, Jain N, Sasaki K, Daver N, Pemmaraju N, Khoury JD, Jorgensen J, Alvarado Y, Konopleva M, Garcia-Manero G, Kadia T, Yilmaz M, Bortakhur G, Burger J, Kornblau S, Wierda W, DiNardo C, Ferrajoli A, Jacob J, Garris R, O'Brien S, Jabbour E. Inotuzumab ozogamicin in combination with low-intensity chemotherapy for older patients with Philadelphia chromosome-negative acute lymphoblastic leukaemia: a single-arm, phase 2 study. Lancet Oncol. 2018 Feb;19(2):240-248. doi: 10.1016/S1470-2045(18)30011-1. Epub 2018 Jan 16. PMID 29352703
- [Derived] Jabbour E, Ravandi F, Kebriaei P, Huang X, Short NJ, Thomas D, Sasaki K, Rytting M, Jain N, Konopleva M, Garcia-Manero G, Champlin R, Marin D, Kadia T, Cortes J, Estrov Z, Takahashi K, Patel Y, Khouri MR, Jacob J, Garris R, O'Brien S, Kantarjian H. Salvage Chemoimmunotherapy With Inotuzumab Ozogamicin Combined With Mini-Hyper-CVD for Patients With Relapsed or Refractory Philadelphia Chromosome-Negative Acute Lymphoblastic Leukemia: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Feb 1;4(2):230-234. doi: 10.1001/jamaoncol.2017.2380. PMID 28859185
- See also: MD Anderson Cancer Center — http://www.mdanderson.org